CLINICAL TRIAL: NCT04376346
Title: Preventing Alcohol Exposed Pregnancy Among Urban Native Young Women: Mobile CHOICES
Acronym: WYSE CHOICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-0574; R01AA025603 (NIH)
Record Dates: First submitted 2020-04-14; First posted 2020-05-06 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Alcohol Exposed Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants in the intervention arm will complete the AIY-C curriculum that has been translated for mHealth delivery. This includes completing various activities such as completing their own risk assessment when it comes to AEP and setting goals for themselves.
  Interventions: Behavioral: Native WYSE CHOICES
- Control Arm (No Intervention): Participants in the control arm will complete activities that are carefully designed under different topics than the intervention arm. In this regard, participants will complete various activities such as quizzes, interactive games and videos. The investigators will ensure that participants in both arms will spend similar time on completing the activities.

INTERVENTIONS:
Behavioral: Native WYSE CHOICES — Native WYSE (Women, Young, Strong, and Empowered) CHOICES (Changing High-risk alcohOl use and Increasing Contraception Effectiveness Study) is an alcohol-exposed pregnancy prevention program that translates CHOICES, an evidence-based targeted intervention, into an mHealth universal intervention for young urban American Indian/Alaska Native (AI/AN) women ages 16-20.
  Arms: Intervention Arm

SUMMARY:
Fetal Alcohol Syndrome Disorders (FASD) result in lifelong disability and are a leading cause of preventable birth defects in the US. Urban American Indian and Alaska Native (AIAN) young women are at high risk for alcohol exposed pregnancies (AEPs) which can cause FASD. In this project, the inverstigators will test the effectiveness of a culturally adapted mobile health intervention to prevent AEP, using social media to recruit AIAN young women from urban centers across the nation.

DETAILED DESCRIPTION:
The proposed project builds on a prior NIAAA-funded project which used intensive community-based participatory research (CBPR) methods to adapt CHOICES, an evidence-based brief alcohol-exposed pregnancy (AEP) prevention intervention supported by the CDC, to American Indian Youth CHOICES (AIY-C). AIY-C contains features that make it highly amenable to mHealth approaches, including a framework for integrating diverse cultural teachings, few modules of short duration, and concrete opportunities for goal-setting and achievement. Innovative for this population is the plan to recruit young AIAN women from major urban areas in the US through social media-and to deliver AIY-C via mobile devices, increasingly ubiquitous among AIAN young adults. While social media recruitment and mHealth interventions are not new, only very recently have they been used with AIAN populations. The investigators will partner with urban AIAN organizations to guide us through social media recruitment strategies, mHealth intervention translation and implementation, and evaluation in urban AIAN settings. The investigators propose 3 specific aims: (1) Develop and pilot social-media-based recruitment strategies for urban AIAN young women; (2) translate AIY-C for mHealth delivery through an iterative and theoretically driven process and pilot the developed translated mHealth AIY-C intervention; and (3) recruit 700 (final N=525) urban AIAN young women using identified social media strategies, and conduct an RCT to rigorously evaluate the effectiveness of the mHealth translation of AIY-C for preventing AEP and FASD.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as American Indian or Alaska Native (AIAN)
* Biologically female
* 16-20 years old
* Not pregnant
* Not living in tribal reservation or in an Alaska Native Village
* Live in an urban area that is at least 50,000 in population
* Not breastfeeding
* Has an email account
* Has a smart phone

Exclusion Criteria:

* Age 15 or younger, and 21 or older
* Biologically male
* Not AIAN
* Pregnant or breastfeeding women
* People who live on a tribal land or in communities with less than 50,000 in population
* Reside in the state of Alaska (until study obtains local IRB approval)

Ages: 16 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 439 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Kaufman, PhD, Principal Investigator — University of Colorado, Denver; Michelle Sarche, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado- Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reed ND, Sarche M, Shrestha U, Bull S, Howley CT, Shangreau C, Asdigian NL, Vossberg RL, Leon JS, Kaufman CE. Creating a Virtual Indigenist Community-Based Participatory Approach: Lessons Learned from Centering Urban Native Young Women in Research. Advers Resil Sci. 2023 Dec;4(4):423-433. doi: 10.1007/s42844-023-00114-z. Epub 2023 Sep 30. PMID 40766111
- [Derived] Reed ND, Bull S, Shrestha U, Sarche M, Kaufman CE. Combating Fraudulent Participation in Urban American Indian and Alaska Native Virtual Health Research: Protocol for Increasing Data Integrity in Online Research (PRIOR). JMIR Res Protoc. 2024 Jun 13;13:e52281. doi: 10.2196/52281. PMID 38869930

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All eligible participants who signed an informed consent completed a baseline survey (online). Once the survey was complete, participants downloaded a mobile app. Upon opening the app they were randomly assigned to either the intervention or control arm, both available within the same app.
  All participants enrolled at baseline are invited to participate in each follow-up survey, regardless of participation status of a previous follow-up survey.
Period: 1 Month Follow up
Arm/Group | Intervention Arm | Control Arm
Started | 218 | 221
Completed | 159 | 166
Not Completed | 59 | 55
Period: 6 Month Follow up
Arm/Group | Intervention Arm | Control Arm
Started | 218 | 221
Completed (All participants enrolled at baseline are invited to participate in each follow-up survey, regardless of participation status of a previous follow-up survey.) | 157 | 157
Not Completed | 61 | 64
Period: 12 Month Follow up
Arm/Group | Intervention Arm | Control Arm
Started | 218 | 221
Completed (All participants enrolled at baseline are invited to participate in each follow-up survey, regardless of participation status of a previous follow-up survey.) | 156 | 164
Not Completed | 62 | 57

BASELINE CHARACTERISTICS:
Population: Participants could not answer any question (per our IRB requirement). Thus, not all participants answered all questions on the baseline survey. Also, all baseline participants were invited to completed a follow-up survey at 1 month; they were also invited to complete surveys at 6, and 12 month follow up periods regardless of whether they completed the prior follow-up survey or not. Thus, some counts across arms will not match the original numbers randomized to each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 218 | 221 | 439
Age, Continuous [Mean (Standard Deviation); unit: year] — Population was defined as those age 16-20
  year | 18.02 (1.39) | 18.16 (1.39) | 18.09 (1.39)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population was defined as females only Population: Participants could choose not to answer any question on this online survey
  Participants
    Female | 194 | 190 | 384
    Trans male | 1 | 1 | 2
    Non-binary | 7 | 17 | 24
    two-spirit | 11 | 8 | 19
    Other/not sure | 3 | 5 | 8
    Missing | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/ethnicity was designed as a "select all that apply"; participants had to select American Indian/Alaska Native as a race to be eligible Population: Participants could choose not to answer any question on this online survey
  Participants
    African American | 12 | 18 | 30
    American Indian/Alaska Native | 218 | 221 | 439
    Asian | 9 | 7 | 16
    Native Hawaiian/Pacific Islander | 2 | 3 | 5
    Hispanic/Latinx | 50 | 66 | 116
    White/Caucasian | 66 | 66 | 132
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Use
Description: Had at least one alcoholic drink in past 30 days (Y/N)
Time Frame: Baseline
Population: Participants could choose not to answer any question on this online survey
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 218 | 221
Participants
  Yes | 86 | 82
  No | 131 | 137
  Missing | 1 | 2

2. Primary Outcome: Alcohol Use
Description: Had at least one alcoholic drink in past 30 days (Y/N)
Time Frame: 1 month
Population: Participants could skip any question on the online survey; we also had attrition at follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 218 | 221
Participants
  Yes | 59 | 60
  No | 93 | 94
  Missing | 66 | 67

3. Primary Outcome: Alcohol Use
Description: Had at least one alcoholic drink in past 30 days (Y/N)
Time Frame: 6 months
Population: Participants could skip any question on the online survey; we also had attrition at follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 218 | 221
Participants
  Yes | 56 | 69
  No | 97 | 86
  Missing | 65 | 66

4. Primary Outcome: Alcohol Use
Description: Had at least one alcoholic drink in past 30 days (Y/N)
Time Frame: 12 months
Population: Participants could skip any question on the online survey; we also had attrition at follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 218 | 221
Participants
  Yes | 71 | 74
  No | 84 | 88
  Missing | 63 | 59

5. Primary Outcome: Effective Contraceptive Use
Description: Effective contraceptive use (including abstinence), measured by past 30-day vaginal sexual abstinence or, if sexually active, 30 day use of effective contraception at intercourse.
Time Frame: Baseline
Population: Participants could skip any question on the online survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 218 | 221
Participants
  Yes | 209 | 197
  No | 9 | 23
  Missing | 0 | 1

6. Primary Outcome: Effective Contraceptive Use
Description: as for outcome 5
Time Frame: 1 months
Population: Participants could skip any question on the online survey; we also had attrition at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 218 | 221
Participants
  Yes | 145 | 143
  No | 7 | 13
  Missing | 66 | 65

7. Primary Outcome: Effective Contraceptive Use
Description: as for outcome 5
Time Frame: 6 months
Population: Participants could skip any question on the online survey; we also had attrition at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 218 | 221
Participants
  Yes | 144 | 140
  No | 10 | 15
  Missing | 64 | 66

8. Primary Outcome: Effective Contraceptive Use
Description: as for outcome 5
Time Frame: 12 months
Population: Participants could skip any question on the online survey; we also had attrition at follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 218 | 221
Participants
  Yes | 146 | 146
  No | 10 | 18
  Missing | 62 | 57

ADVERSE EVENTS:
Time Frame: from enrollment to final follow-up (12 months)
Description: Because this was a virtual, national study (virtually no in-person contact), we assessed events by survey data only.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/218 | 0/221
Serious Adverse Events (participants affected / at risk) | 0/218 | 0/221
Other Adverse Events (participants affected / at risk) | 0/218 | 0/221

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT04376346/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT04376346/ICF_001.pdf